CLINICAL TRIAL: NCT02167217
Title: Phase 2 Historically Controlled Trial of Corticosteroids in Young Boys With Duchenne Muscular Dystrophy
Brief Title: Historically Controlled Trial of Corticosteroids in Young Boys With Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Nationwide Children's Hospital (Other); Northwestern University Feinberg School of Medicine (Other); University of Texas Southwestern Medical Center (Other); University of California, Davis (Other); Nemours Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201308062
Record Dates: First submitted 2014-02-03; First posted 2014-06-19 (Estimated); Results first posted 2018-05-18 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; Corticosteroids; Infants; Young Children; Toddlers
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oral Prednisolone (Experimental): Oral Prednisolone 5mg/kg/ day on two consecutive days, Friday and Saturday with breakfast
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Prednisolone — Prednisolone (5mg per kg) will be taken on two consecutive days, Friday and Saturday mornings each week with breakfast
  Other Names: prednisolone (Morton Grove Pharm.) National Drug Code is 60432-212-08

SUMMARY:
While it has been known for many years that corticosteroid use benefits boys with Duchenne Muscular dystrophy (DMD), most clinicians do not consider treating until after age 3 or 4 years of age. The primary reason for the delay is that daily corticosteroid use has many side effects including short stature, obesity, and osteoporosis. A recent randomized blinded study of weekend oral corticosteroid use over one year showed equal improvement in strength with fewer side effects, particularly as related to growth and cushingoid changes. The investigators will test the efficacy of oral weekend corticosteroid use in infants and young boys with DMD who are under age 30 months. The investigators have demonstrated that the Bayley-III Scales of Infant development shows that infants and young boys in this age group who are untreated decline in abilities when compared to their peers. Here, in this Phase 2 historically controlled trial, the investigators will use these two measures and treat boys at five Muscular Dystrophy Association-DMD centers

DETAILED DESCRIPTION:
Objective. Determine if twice-weekly high dose oral prednisone improves gross motor development in infants and young boys with DMD. The investigators will perform a phase 2 historically controlled trial of oral twice-weekly prednisone (5mg/kg/dose on two consecutive days) in infants and young boys with DMD. Here the investigators propose to study the effect of this therapy in a multicenter trial of boys with DMD who are less than 30 months old at the baseline visit. Each boy will be followed for one year.

Aim 1. Determine if treatment improves gross motor function in infants with DMD over a 6-12-month period as measured by the Bayley-III. The Bayley-III infant score is the primary motor clinical endpoint of this therapeutic trial. Secondary outcomes include fine motor function, speech and language, and social function.

Aim 2. Determine if treatment improves the Adaptive Behavior Subtest of the Bayley-III (ABS) as scored by the infants' primary caregiver. In the study of untreated boys, the primary caregiver noted clear deficits, predominantly related to areas relevant to gross motor function. The ABS Aim 3. Determine if treatment improves performance on the North Star Ambulatory Assessment (NSAA) for those boys who are ambulatory.

Aim 4. Determine if treatment with weekly corticosteroids is tolerated and is safe in boys with DMD who are less than 30 months of age.

Objective 2. Determine if ultrasound of biceps and quadriceps using calibrated backscatter improves in infants and young boys with DMD who are treated with oral high dose weekly corticosteroids. Preliminary data of ultrasound imaging in infants and young boys with DMD demonstrate progressive structural damage as measured by calibrated backscatter. The ultrasound studies will be limited to the infants and boys who will enroll at the primary site (Washington University) where Dr. Craig Zaidman has the equipment and expertise to accomplish this aim.

Objective 3. Determine if caregiver burden changes with treatment of infants and young boys with DMD. Preliminary data from questionnaires suggests the caregiver burden for the primary caregiver of untreated infant and young boys with DMD is minimal. Assessment of this with in this trial will allow us to discern if this changes with a therapeutic trial.

ELIGIBILITY:
Inclusion Criteria:

1. Appropriate degree of weakness for age, creatine kinase greater than 20 times the upper limit of normal, and genetic mutation known to be causative for Duchenne muscular dystrophy .
2. Appropriate degree of weakness for age, creatine kinase greater than 20 times the upper limit of normal and genetic or biopsy confirmation of Duchenne muscular dystrophy in a primary relative (e.g. brother or maternal uncle).
3. De-identified, genetic studies will be reviewed by collaborator Kevin Flanigan, MD prior to enrollment of subjects.
4. Age at entry: one month through 30 months.

Exclusion Criteria:

* Prior treatment with corticosteroids

Ages: 1 Month to 30 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2014-04-17 (Actual); Primary Completion 2017-02-22 (Actual); Study Completion 2017-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Connolly, MD, Principal Investigator — Washington University School of Medicine
Locations (6):
- United States (6):
  - University of California Davis, Sacramento, California
  - Nemours Hospital, Orlando, Florida
  - Laurie Children's Hospital Of Chicago, Chicago, Illinois
  - Washington University in Saint Louis, St Louis, Missouri
  - Research Institute Center for Gene Therapy at Nationwide Children's Hospital, Columbus, Ohio
  - University of Texas South Western Medical Center of Dallas, Dallas, Texas

REFERENCES:
- [Background] Connolly AM, Florence JM, Cradock MM, Malkus EC, Schierbecker JR, Siener CA, Wulf CO, Anand P, Golumbek PT, Zaidman CM, Philip Miller J, Lowes LP, Alfano LN, Viollet-Callendret L, Flanigan KM, Mendell JR, McDonald CM, Goude E, Johnson L, Nicorici A, Karachunski PI, Day JW, Dalton JC, Farber JM, Buser KK, Darras BT, Kang PB, Riley SO, Shriber E, Parad R, Bushby K, Eagle M; MDA DMD Clinical Research Network. Motor and cognitive assessment of infants and young boys with Duchenne Muscular Dystrophy: results from the Muscular Dystrophy Association DMD Clinical Research Network. Neuromuscul Disord. 2013 Jul;23(7):529-39. doi: 10.1016/j.nmd.2013.04.005. Epub 2013 May 28. PMID 23726376
- [Background] Connolly AM, Schierbecker J, Renna R, Florence J. High dose weekly oral prednisone improves strength in boys with Duchenne muscular dystrophy. Neuromuscul Disord. 2002 Dec;12(10):917-25. doi: 10.1016/s0960-8966(02)00180-3. PMID 12467746
- [Background] Escolar DM, Hache LP, Clemens PR, Cnaan A, McDonald CM, Viswanathan V, Kornberg AJ, Bertorini TE, Nevo Y, Lotze T, Pestronk A, Ryan MM, Monasterio E, Day JW, Zimmerman A, Arrieta A, Henricson E, Mayhew J, Florence J, Hu F, Connolly AM. Randomized, blinded trial of weekend vs daily prednisone in Duchenne muscular dystrophy. Neurology. 2011 Aug 2;77(5):444-52. doi: 10.1212/WNL.0b013e318227b164. Epub 2011 Jul 13. PMID 21753160
- [Derived] Connolly AM, Zaidman CM, Golumbek PT, Cradock MM, Flanigan KM, Kuntz NL, Finkel RS, McDonald CM, Iannaccone ST, Anand P, Siener CA, Florence JM, Lowes LP, Alfano LN, Johnson LB, Nicorici A, Nelson LL, Mendell JR; MDA DMD Clinical Research Network. Twice-weekly glucocorticosteroids in infants and young boys with Duchenne muscular dystrophy. Muscle Nerve. 2019 Jun;59(6):650-657. doi: 10.1002/mus.26441. Epub 2019 Feb 23. PMID 30706490

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Prednisolone: Oral Prednisolone 5mg/kg/ day on two consecutive days, Friday and Saturday with breakfast
  Prednisolone: Prednisolone (5mg per kg )will be taken on two consecutive days, Friday and Saturday mornings each week with breakfast
Period: Overall Study
Arm/Group | Oral Prednisolone
Started | 25
Completed | 23
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Two of the 25 dropped out of study. One was lost to followup within a few months and the second discontinued the study after 6 months.
Groups:
- Oral Prednisolone: Oral Prednisolone 5mg/kg/ day on two consecutive days, Friday and Saturday with breakfast
  Prednisolone: Prednisolone (5mg per kg )will be taken on two consecutive days, Friday and Saturday mornings each week with breakfast
  Twenty-five steroid naïve boys four to 30 months of age with genetically confirmed Duchenne Muscular Dystrophy (DMD) were enrolled. 25 infants and boys were enrolled and 23 completed the study. One boy was lost to follow-up and one discontinued treatment after six months secondary to side effects.
Arm/Group | Oral Prednisolone
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants] — Population: The analysis population does not include the two who dropped out.
  Participants
    number analyzed (Participants) | 23
    <=18 years | 23
    Between 18 and 65 years | 0
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The 23 analyzed does not include the two who dropped out.
  years
    number analyzed (Participants) | 23
    (all) | 1.5 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The number analyzed does not include the two who dropped out. See above.
  Participants
    number analyzed (Participants) | 23
    Female | 0
    Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 22
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants] — Population: The number analyzed does not include the two who dropped out
  Participants
    United States: number analyzed (Participants) | 23
    United States | 23
Bayley III Gross Motor Scaled Score [Mean (Standard Deviation); unit: units on a scale] — This scale is normed to typically developing children where at any age a child's expected score is 10 +/-3. This scale assesses gross motor function including sitting, standing and walking. Population: The number analyzed does not include the two who dropped out.
  units on a scale
    number analyzed (Participants) | 23
    (all) | 4.2 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Bayley III Gross Motor Scaled Score (Change From Baseline to 12 Month)
Description: Bayley III Gross Motor Scaled Score measures motor development. This is normed for typically developing children and follow a bell shaped curve. The scale has mean of 10 +/-3 for children at all ages and is bell shaped. Therefore the two standard deviation range is 16 to 4 with higher values indicated better performance. Lower values have been shown to be common in boys with DMD and it this study the baseline average score was 4.2.
Time Frame: One year
Population: We analyzed the change in the gross motor score after one year. An increase indicates improvement compared to peers
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oral Prednisolone
Number analyzed (Participants) | 23
units on a scale | 4.8 (2.3)

ADVERSE EVENTS:
Time Frame: Data for adverse event were collected over one year.
Description: 60 adverse events (AEs) were reported; 15 were possibly or probably related to medication. There were no severe AEs.
Arm/Group | Oral Prednisolone
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 22/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Prednisolone (N=25)
irritability (Nervous system disorders) | 4 (7) — Irritability occurred 10 times in 4 children.
Upper Respiratory Track Infection (Respiratory, thoracic and mediastinal disorders) | 14 (17)
Gastroenteritis (Gastrointestinal disorders) | 5 (5)
Ear Infection (Infections and infestations) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Fever (General disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/17/NCT02167217/SAP_000.pdf
  • Study Protocol (2013-10-02): https://cdn.clinicaltrials.gov/large-docs/17/NCT02167217/Prot_002.pdf